CLINICAL TRIAL: NCT00735709
Title: A Randomized, Double-blind, Parallel-Group, Placebo-Controlled, Fixed-Dose Study Comparing the Efficacy and Safety of 3 Doses of Lu AA21004 in Acute Treatment of Adults With Major Depressive Disorder
Brief Title: Efficacy Study of Vortioxetine (Lu AA21004) in Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LuAA21004_305; 2008-001580-11 (EudraCT Number); U1111-1114-0326 (Registry Identifier: WHO)
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Depressive Disorder; Mood Disorder; Mental Disorder; Melancholia, Involutional; Paraphrenia, Involutional; Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder; Mood Disorders; Mental Disorders | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vortioxetine 1 mg (Experimental): Vortioxetine 1 mg, encapsulated tablets, orally, once daily for up 8 weeks.
  Interventions: Drug: Vortioxetine
- Vortioxetine 5 mg (Experimental): Vortioxetine 5 mg, encapsulated tablets, orally, once daily for up 8 weeks.
  Interventions: Drug: Vortioxetine
- Vortioxetine 10 mg (Experimental): Vortioxetine 10 mg, encapsulated tablets, orally, once daily for up 8 weeks.
  Interventions: Drug: Vortioxetine
- Placebo (Placebo Comparator): Vortioxetine placebo-matching capsules, orally, once daily for up to 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine — Encapsulated immediate-release vortioxetine tablets
  Other Names: Lu AA21004; Brintellix®
  Arms: Vortioxetine 1 mg; Vortioxetine 10 mg; Vortioxetine 5 mg
Drug: Placebo — Vortioxetine placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of vortioxetine, once daily (QD), in patients with Major Depressive Disorder.

DETAILED DESCRIPTION:
The drug that was tested in this study is called vortioxetine. Vortioxetine is being tested to treat depression in adults who have major depressive disorder (MDD). This study looked at MDD relief in people who took varying dosages of vortioxetine.

The study enrolled 560 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the four treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Vortioxetine 1 mg
* Vortioxetine 5 mg
* Vortioxetine 10 mg
* Placebo (dummy inactive pill) - this was a capsule that looked like the study drug but had no active ingredient.

All participants were asked to take one capsule at the same time each day throughout the study.

This multi-centre trial was conducted in Europe, Asia, Australia, and South Africa. The overall time to participate in this study was up to 14 weeks. Participants made 7 visits to the clinic, and were contacted by telephone 4 weeks after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Has a primary diagnosis of major depressive episode according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria.
* The reported duration of the current major depressive episode is at least 3 months.
* Has a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≥26.
* A male or a female of childbearing potential who is sexually active agrees to use adequate contraception from Screening throughout the duration of the study and for 1 month after the last dose of study medication.

Exclusion Criteria:

* Has 1 or more the following:

  * Any current psychiatric disorder other than major depressive disorder as defined in the DSM-IV-TR.
  * Current or past history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
  * Any substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR. (must have negative urine drug screen prior to Baseline).
  * Presence or history of a clinically significant neurological disorder (including epilepsy).
  * Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
* Has a significant risk of suicide according to the investigator's opinion or has a score ≥5 on item 10 (suicidal thoughts) of the Montgomery Åsberg Depression Rating Scale, or has made a suicide attempt in the previous 6 months.
* Currently receiving formal cognitive or behavioral therapy, systematic psychotherapy, or plans to initiate such therapy during the study.
* Has a clinically significant unstable illness.
* Has previously failed to respond to adequate treatment with selective serotonin reuptake inhibitors and/or serotonin-norepinephrine reuptake inhibitors.
* Has received electroconvulsive therapy within 6 months prior to Screening.
* Has an alanine aminotransferase, aspartate aminotransferase, or total bilirubin level > 1.5 times the upper limit of normal.
* Has a serum creatinine of > 1.5 × upper limit of normal.
* Has a previous history of cancer that had been in remission for less than 5 years.
* Has thyroid stimulating hormone value outside the normal range.
* Has an abnormal electrocardiogram.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (48):
- Australia (2):
  - Elizabeth Vale
  - Southport
- Czechia (3):
  - Litoměřice
  - Lnáře
  - Prague
- France (3):
  - Bully-les-Mines
  - Marseille
  - Strasbourg
- Germany (10):
  - Bochum
  - Chemnitz
  - Dillingen
  - Hüttenberg
  - Leipzig
  - München
  - Nuremberg
  - Osnabrück
  - Rodgau
  - Westerstede
- Latvia (4):
  - Leipaja
  - Riga
  - Sigulda
  - Strenči
- Vilnius, Lithuania
- Kuala Lumpur, Malaysia
- Wildervank, Netherlands
- Poland (5):
  - Bialystok
  - Leszno
  - Skórzewo
  - Torun
  - Tuszyn
- Russia (5):
  - Moscow
  - Saint Petersburg
  - Stavropol
  - Tomsk
  - Veliky Novgorod
- South Africa (3):
  - Durban
  - Noordheuwel
  - Pretoria
- South Korea (3):
  - Bucheon-si
  - Namdong-gu
  - Seoul
- Lin-Yan District, Taiwan
- Ukraine (4):
  - Dnipro
  - Kharkiv
  - Luhansk
  - Simferopol
- United Kingdom (2):
  - Bath
  - Bolton

REFERENCES:
- [Background] Henigsberg N, Mahableshwarkar AR, Jacobsen P, Chen Y, Thase ME. A randomized, double-blind, placebo-controlled 8-week trial of the efficacy and tolerability of multiple doses of Lu AA21004 in adults with major depressive disorder. J Clin Psychiatry. 2012 Jul;73(7):953-9. doi: 10.4088/JCP.11m07470. PMID 22901346
- [Derived] McIntyre RS, Florea I, Tonnoir B, Loft H, Lam RW, Christensen MC. Efficacy of Vortioxetine on Cognitive Functioning in Working Patients With Major Depressive Disorder. J Clin Psychiatry. 2017 Jan;78(1):115-121. doi: 10.4088/JCP.16m10744. PMID 27780334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 51 investigative sites in Australia, Croatia, France, Germany, Latvia, Lithuania, Malaysia, Netherlands, Poland, Republic of Korea, Russia, South Africa, Taiwan, and Ukraine from 14 August 2008 to 13 August 2009.
Pre-assignment Details: Participants with a diagnosis of major depressive disorder were randomized equally in 1 of 4 treatment groups, once daily placebo, 1 mg, 5 mg, or 10 mg vortioxetine.
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Started | 140 | 140 | 140 | 140
Treated | 140 | 140 | 140 | 139
Completed | 127 | 127 | 129 | 122
Not Completed | 13 | 13 | 11 | 18
Not completed — Adverse Event | 2 | 3 | 1 | 5
Not completed — Lack of Efficacy | 8 | 4 | 2 | 3
Not completed — Noncompliance | 0 | 0 | 1 | 0
Not completed — Protocol deviations | 1 | 2 | 1 | 1
Not completed — Voluntary Withdrawal | 1 | 3 | 5 | 7
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Excluded medication | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Total
Number analyzed (Participants) | 140 | 140 | 140 | 140 | 560
Age Continuous [Mean (Standard Deviation); unit: years] | 46.4 (12.26) | 45.4 (11.89) | 47.3 (11.95) | 46.4 (12.27) | 46.4 (12.08)
Age, Customized [Number; unit: participants]
  ≤55 years | 103 | 110 | 102 | 107 | 422
  >55 years | 37 | 30 | 38 | 33 | 138
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 93 | 87 | 85 | 351
  Male | 54 | 47 | 53 | 55 | 209
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 120 | 129 | 120 | 114 | 483
  Black | 5 | 1 | 2 | 2 | 10
  Asian | 14 | 8 | 17 | 23 | 62
  Other | 1 | 2 | 1 | 1 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 3 | 0 | 0 | 1 | 4
  Non-Hispanic/Non-Latino | 137 | 140 | 140 | 139 | 556
Region of Enrollment [Number; unit: participants]
  Australia | 0 | 3 | 0 | 1 | 4
  Croatia | 2 | 5 | 5 | 1 | 13
  France | 5 | 2 | 1 | 5 | 13
  Germany | 63 | 50 | 64 | 56 | 233
  Latvia | 5 | 8 | 9 | 5 | 27
  Lithuania | 4 | 4 | 2 | 3 | 13
  Malaysia | 7 | 3 | 6 | 6 | 22
  Netherlands | 0 | 3 | 3 | 1 | 7
  Poland | 20 | 16 | 15 | 11 | 62
  Republic of Korea | 7 | 5 | 9 | 14 | 35
  Russia | 12 | 20 | 9 | 20 | 61
  South Africa | 5 | 6 | 5 | 3 | 19
  Taiwan | 0 | 0 | 1 | 3 | 4
  Ukraine | 10 | 15 | 11 | 11 | 47
Weight [Mean (Standard Deviation); unit: kg] | 75.18 (14.924) | 75.63 (17.276) | 75.41 (17.022) | 74.58 (15.190) | 75.20 (16.099)
Height [Mean (Standard Deviation); unit: cm] | 168.70 (8.907) | 168.56 (8.264) | 168.56 (9.126) | 168.70 (10.209) | 168.63 (9.129)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.36 (4.615) | 26.53 (5.380) | 26.41 (5.065) | 26.16 (4.612) | 26.36 (4.917)
Smoking Classification [Number; unit: participants]
  Never smoked | 88 | 74 | 88 | 79 | 329
  Current smoker | 34 | 54 | 33 | 41 | 162
  Ex-smoker | 18 | 12 | 19 | 20 | 69
Alcohol Consumption [Number; unit: participants]
  Never | 53 | 51 | 56 | 54 | 214
  Once monthly or less often | 57 | 60 | 59 | 51 | 227
  Once per week | 16 | 13 | 9 | 16 | 54
  2-to-6 times/week | 5 | 11 | 7 | 12 | 35
  Daily | 9 | 5 | 9 | 7 | 30
24-item Hamilton Depression Scale total score [Mean (Standard Deviation); unit: scores on a scale] — The 24-item Hamilton Depression Scale (HAM-D24) is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74, where a higher score indicates a greater depressive state.
  scores on a scale | 32.7 (4.40) | 32.5 (5.13) | 32.1 (5.04) | 33.1 (4.77) | 32.6 (4.84)
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 30.6 (2.89) | 30.4 (3.01) | 30.6 (2.83) | 31.6 (3.83) | 30.8 (3.19)
Hamilton Anxiety Scale total score [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety.
  scores on a scale | 19.7 (7.07) | 20.0 (6.41) | 19.4 (6.77) | 21.1 (7.39) | 20.0 (6.93)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  scores on a scale | 4.8 (0.80) | 4.7 (0.73) | 4.8 (0.73) | 4.9 (0.76) | 4.8 (0.76)
Hospital Anxiety and Depression (HAD) - Anxiety subscale [Mean (Standard Deviation); unit: scores on a scale] — The HAD-anxiety subscale is completed by the participant and measures anxiety, including anxious mood, restlessness, anxious thoughts, and panic attacks. The subscale is made up of 7 items that are assessed on a scale from 0 (no anxiety) to 3 (severe feeling of anxiety). Participants are required to indicate the response which most accurately reflects the way they have felt over the last few days. Scores are summed and range from 0 to 21 (maximal severity).
  scores on a scale | 11.2 (3.99) | 11.2 (3.83) | 11.6 (4.02) | 11.7 (3.97) | 11.4 (3.95)
Hospital Anxiety and Depression - Depression subscale [Mean (Standard Deviation); unit: scores on a scale] — The HAD - Depression subscale is completed by the participant and measures depression, focusing on the state of lost interest and diminished pleasure response. The subscale is made up of 7 items that are assessed on a scale from 0 (no depression) to 3 (severe feeling of depression). Participants are required to indicate the response which most accurately reflects the way they have felt over the last few days. The item scores are summed and the total subscore ranges from 0 to 21 (maximal severity).
  scores on a scale | 13.7 (4.33) | 13.8 (3.88) | 13.4 (4.02) | 13.8 (3.71) | 13.7 (3.99)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 24-item Hamilton Depression Scale Total Score At Week 8
Description: The 24-item Hamilton Depression Scale (HAM-D24) is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score range is from 0 to 74 where a higher score indicates a greater depressive state. Least squares (LS) means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Week 8
Population: The full analysis set (FAS) included all patients who were randomized, received at least 1 dose of study drug, and had at least 1 post-baseline value for assessment of primary efficacy. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 128 | 124 | 129 | 122
scores on a scale | -11.30 (0.738) | -14.82 (0.745) | -15.42 (0.743) | -16.23 (0.755)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; All statistical tests were 2-sided with the estimated P-values at the 5% level of significance. To control for multiplicity, a pre-specified sequential testing procedure was applied to compare 10 mg and 5 mg vortioxetine to placebo; as soon as an endpoint was non-significant at 0.05, the testing procedure stopped for all subsequent endpoints; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — Pre-specified sequential statistical testing procedure indicates that when p-value <0.05, hierarchical testing continues; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -4.93, 95% CI 2-sided [-6.99 to -2.86]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — Hierarchical testing stopped at SDS total score at Week 8 in the testing sequence, a nominal p-value is provided; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -4.12, 95% CI 2-sided [-6.17 to -2.08]
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 1 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — This treatment arm is not in the testing sequence, a nominal p-value is provided; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -3.52, 95% CI 2-sided [-5.57 to -1.47]

2. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 8
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 94 | 90 | 97 | 83
scores on a scale | -6.54 (0.716) | -6.58 (0.729) | -7.65 (0.713) | -8.08 (0.756)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.135, Mixed model repeated measurements — Pre-specified sequential statistical testing procedure indicates that when p-value >0.05, hierarchical testing stops and for subsequent endpoints in the sequence a nominal p-value is provided; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -1.54, 95% CI 2-sided [-3.56 to 0.48]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.263, Mixed model repeated measurements; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -1.11, 95% CI 2-sided [-3.07 to 0.84]
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 1 mg; Test type: Superiority or Other; p = 0.963, Mixed model repeated measurements; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -0.05, 95% CI 2-sided [-2.03 to 1.94]

3. Secondary Outcome: Clinical Global Impression Scale-Global Improvement at Week 8
Description: The Clinical Global Impression - Global Improvement scale assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 128 | 124 | 129 | 122
scores on a scale | 2.84 (0.089) | 2.37 (0.090) | 2.37 (0.089) | 2.29 (0.091)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p < 0.001, Mixed model repeated measurements; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -0.55, 95% CI 2-sided [-0.80 to -0.30]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.001, Mixed model repeated measurements; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -0.47, 95% CI 2-sided [-0.71 to -0.22]
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 1 mg; Test type: Superiority or Other; p < 0.001, Mixed model repeated measurements; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -0.47, 95% CI 2-sided [-0.72 to -0.23]

4. Secondary Outcome: Percentage of Responders in HAM-D24 Total Score at Week 8
Description: A responder is defined as a participant with a ≥50% decrease from Baseline in HAM-D24 total score. The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74, where a higher score indicates a greater depressive state.
Time Frame: Baseline and Week 8
Population: Full analysis set; last observation carried forward (LOCF) was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
percentage of participants | 23.0 | 47.5 | 45.3 | 49.6
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Regression with explanatory variables for treatment and Baseline HAM-D24 score; Odds Ratio (OR) = 3.348, 95% CI 2-sided [1.995 to 5.618] — Odds ratio versus placebo
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Regression with explanatory variables for treatment and Baseline HAM-D24 score; Odds Ratio (OR) = 2.739, 95% CI 2-sided [1.631 to 4.598] — Odds ratio versus placebo
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 1 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Regression with explanatory variables for treatment and Baseline HAM-D24 score; Odds Ratio (OR) = 3.018, 95% CI 2-sided [1.799 to 5.063] — Odds ratio versus placebo

5. Secondary Outcome: Change From Baseline in HAM-D24 Total Score at Week 8 in Participants With Baseline HAM-A Score ≥20
Description: The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74 where a higher score indicates a greater depressive state. The Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (symptoms absent) to 56 (severe symptoms). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline to Week 8
Population: Full analysis set patients with a HAM-A Baseline score ≥ 20. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 62 | 65 | 57 | 65
scores on a scale | -11.02 (1.017) | -15.16 (0.991) | -15.50 (1.063) | -15.61 (0.984)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.001, Mixed model for repeated measurements; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -4.59, 95% CI 2-sided [-7.34 to -1.84]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.002, Mixed model for repeated measurements; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -4.47, 95% CI 2-sided [-7.32 to -1.62]
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 1 mg; Test type: Superiority or Other; p = 0.004, Mixed model for repeated measurements; P-values are from an MMRM model with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis; LS Mean Difference = -4.13, 95% CI 2-sided [-6.90 to -1.37]

6. Secondary Outcome: Percentage of Participants in MADRS Remission at Week 8
Description: Remission is defined as a participant with a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≤10. The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement.
Time Frame: Week 8
Population: Full analysis set; LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
percentage of participants | 16.5 | 25.9 | 28.8 | 26.6
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.026, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline MADRS score; Odds Ratio (OR) = 1.951, 95% CI 2-sided [1.082 to 3.517]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.015, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline MADRS score; Odds Ratio (OR) = 2.056, 95% CI 2-sided [1.150 to 3.673]
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 1 mg; Test type: Superiority or Other; p = 0.062, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline MADRS score; Odds Ratio (OR) = 1.753, 95% CI 2-sided [0.973 to 3.158]

7. Secondary Outcome: Change From Baseline in the 24-item Hamilton Depression Scale Total Score at Other Weeks Assessed
Description: The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score range is from 0 to 74 where a higher score indicates a greater depressive state. LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 1, 2, 4 and 6
Population: Full analysis set with available data at Baseline. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
scores on a scale
  Week 1 (n=139, 137, 138, 138) | -3.47 (0.321) | -2.81 (0.323) | -3.20 (0.322) | -3.20 (0.321)
  Week 2 (n=138, 138, 135, 135) | -5.66 (0.485) | -7.27 (0.485) | -7.27 (0.490) | -7.42 (0.489)
  Week 4 (n=135, 133, 135, 127) | -8.42 (0.634) | -11.09 (0.637) | -11.00 (0.639) | -11.88 (0.646)
  Week 6 (n=134, 130, 129, 126) | -10.23 (0.690) | -13.35 (0.695) | -13.67 (0.697) | -15.22 (0.705)

8. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Other Weeks Assessed
Description: as for outcome 2
Time Frame: Baseline and Weeks 1, 2 and 6
Population: Full analysis set with available SDS Total Score data at Baseline. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 104 | 103 | 106 | 99
scores on a scale
  Week 1 (n=104, 101, 105, 97) | -1.22 (0.392) | -1.13 (0.399) | -1.78 (0.393) | -1.43 (0.403)
  Week 2 (n=102, 101, 100, 96) | -2.53 (0.507) | -3.44 (0.511) | -4.14 (0.512) | -3.40 (0.521)
  Week 6 (n=99, 97, 97, 88) | -5.95 (0.672) | -5.69 (0.681) | -6.92 (0.678) | -8.27 (0.707)

9. Secondary Outcome: Clinical Global Impression Scale-Global Improvement at Other Weeks Assessed
Description: The Clinical Global Impression - global improvement assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 1, 2, 4 and 6
Population: Full analysis set with available CGI-S data at Baseline. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
scores on a scale
  Week 1 (n=139, 137, 138, 138) | 3.65 (0.053) | 3.71 (0.054) | 3.67 (0.053) | 3.64 (0.053)
  Week 2 (n=138, 138, 135, 135) | 3.40 (0.069) | 3.16 (0.070) | 3.19 (0.070) | 3.23 (0.070)
  Week 4 (n=135, 133, 135, 127) | 3.03 (0.082) | 2.69 (0.083) | 2.82 (0.083) | 2.78 (0.084)
  Week 6 (n=134, 130, 129, 126) | 2.95 (0.087) | 2.48 (0.088) | 2.50 (0.088) | 2.37 (0.089)

10. Secondary Outcome: Percentage of Responders in HAM-D24 Total Score at Other Weeks Assessed
Description: as for outcome 4
Time Frame: Baseline and Weeks 1, 2, 4 and 6
Population: Full analysis set with available data at Week 1; Last observation carried forward (LOCF) was used for other time points. "n" indicates the number of patients included in the analysis at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
percentage of participants
  Week 1 (n=139, 137, 138, 138) | 0.7 | 0.7 | 0.7 | 1.4
  Week 2 (n=139, 139, 139, 139) | 5.0 | 7.9 | 7.2 | 8.6
  Week 4 (n=139, 139, 139, 139) | 18.0 | 27.3 | 24.5 | 26.6
  Week 6 (n=139, 139, 139, 139) | 23.7 | 38.1 | 36.0 | 43.9

11. Secondary Outcome: Change From Baseline in HAM-D24 Total Score at Other Weeks Assessed in Participants With a Baseline HAM-A Score ≥20
Description: The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score range from 0 to 74 where a higher score indicates a greater depressive state. The Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (symptoms absent) to 56 (symptoms severe). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 1, 2, 4 and 6
Population: Full analysis set patients with a HAM-A Baseline score ≥20 and with available data at Baseline. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 66 | 70 | 62 | 75
scores on a scale
  Week 1 (n=66, 70, 62, 75) | -3.79 (0.473) | -2.94 (0.463) | -3.55 (0.491) | -3.19 (0.447)
  Week 2 (n=65, 70, 59, 72) | -5.76 (0.637) | -7.21 (0.618) | -6.58 (0.667) | -7.74 (0.607)
  Week 4 (n=64, 68, 60, 69) | -8.56 (0.874) | -11.41 (0.850) | -10.20 (0.910) | -12.06 (0.841)
  Week 6 (n=64, 67, 57, 68) | -10.25 (0.958) | -13.68 (0.932) | -13.23 (1.002) | -15.10 (0.923)

12. Secondary Outcome: Percentage of Participants in MADRS Remission at Other Weeks Assessed
Description: as for outcome 6
Time Frame: Weeks 1, 2, 4 and 6
Population: Full analysis set with available data at Week 1; Last observation carried forward was used for other time points.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
percentage of participants
  Week 1 (n=139, 137, 138, 138) | 0.7 | 0.7 | 0 | 0
  Week 2 (n=139, 139, 139, 139) | 2.2 | 2.2 | 1.4 | 1.4
  Week 4 (n=139, 139, 139, 139) | 6.5 | 11.5 | 11.5 | 10.8
  Week 6 (n=139, 139, 139, 139) | 10.1 | 20.1 | 20.9 | 22.3

13. Secondary Outcome: Percentage of Participants With a Sustained Response in HAM-D24 Total Score
Description: A sustained response is defined as a ≥20% decrease from Baseline in HAM-D24 total score obtained at Week 1 and sustained through Week 7 and at least 50% decrease from Baseline at Week 8.
Time Frame: From Baseline through Week 8
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
percentage of participants | 10.1 | 9.4 | 10.1 | 10.8

14. Secondary Outcome: Change From Baseline in Montgomery Åsberg Depression Rating Scale (MADRS) Total Score at Each Week
Description: The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). A decrease in the total score or on individual items indicates improvement. LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 1, 2, 4, 6, and 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
scores on a scale
  Week 1 (n=139, 137, 138, 138) | -2.90 (0.324) | -2.55 (0.326) | -2.66 (0.324) | -2.57 (0.328)
  Week 2 (n=138, 138, 135, 135) | -4.92 (0.463) | -6.65 (0.463) | -6.40 (0.467) | -6.51 (0.472)
  Week 4 (n=135, 133, 135, 127) | -7.85 (0.619) | -10.79 (0.622) | -10.30 (0.622) | -10.89 (0.635)
  Week 6 (n=134, 130, 129, 126) | -9.72 (0.675) | -13.16 (0.680) | -13.10 (0.680) | -14.19 (0.694)
  Week 8 (n=128, 124, 129, 122) | -10.91 (0.708) | -14.89 (0.715) | -15.09 (0.712) | -15.65 (0.728)

15. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) Total Score at Each Week Assessed
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 1, 2, 4, 6, and 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
scores on a scale
  Week 1 (n=139, 137, 138, 138) | -1.58 (0.260) | -1.27 (0.261) | -1.41 (0.261) | -1.56 (0.261)
  Week 2 (n=138, 138, 135, 135) | -3.06 (0.343) | -3.72 (0.343) | -3.09 (0.346) | -3.77 (0.347)
  Week 4 (n=135, 133, 135, 127) | -4.54 (0.416) | -5.95 (0.418) | -5.60 (0.418) | -6.11 (0.425)
  Week 6 (n=134, 130, 129, 126) | -5.44 (0.471) | -7.29 (0.475) | -7.21 (0.476) | -8.33 (0.483)
  Week 8 (n=128, 124, 129, 122) | -5.98 (0.498) | -8.08 (0.503) | -8.11 (0.501) | -8.86 (0.511)

16. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Severity of Illness at Each Week Assessed
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 1, 2, 4, 6, and 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
scores on a scale
  Week 1 (n=139, 137, 138, 138) | -0.24 (0.044) | -0.20 (0.045) | -0.22 (0.044) | -0.24 (0.044)
  Week 2 (n=138, 138, 135, 135) | -0.46 (0.062) | -0.58 (0.062) | -0.61 (0.062) | -0.60 (0.062)
  Week 4 (n=135, 133, 135, 127) | -0.75 (0.080) | -1.07 (0.081) | -1.10 (0.081) | -1.06 (0.082)
  Week 6 (n=134, 130, 129, 126) | -0.96 (0.092) | -1.41 (0.093) | -1.38 (0.093) | -1.55 (0.094)
  Week 8 (n=128, 124, 129, 122) | -1.12 (0.101) | -1.50 (0.102) | -1.63 (0.101) | -1.74 (0.103)

17. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression (HAD) Scales at Each Week Assessed
Description: The HAD scale is completed by the participant and comprises two subscales, one measuring depression (focusing on the state of lost interest and diminished pleasure response) and one measuring anxiety (including anxious mood, restlessness, anxious thoughts, panic attacks). Each subscale is made up of 7 items that are assessed on a scale of 0 = no anxiety/depression to 3 = severe feeling of anxiety/depression. Participants are required to indicate the response which most accurately reflects the way they have felt over the last few days. Scores for the depression and anxiety subscales are summed separately and not combined, with each score ranging from 0 to 21 (maximal severity). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis
Time Frame: Baseline and Weeks 1, 4, and 8
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 138
scores on a scale
  Anxiety Scale at Week 1 (n=139, 137, 138, 137) | -0.46 (0.190) | -1.14 (0.190) | -0.87 (0.189) | -0.91 (0.190)
  Anxiety Scale at Week 4 (n=137, 138, 135, 134) | -1.95 (0.277) | -2.83 (0.276) | -2.81 (0.278) | -2.80 (0.279)
  Anxiety Scale at Week 8 (n=129, 129, 127, 122) | -2.55 (0.315) | -3.79 (0.315) | -3.70 (0.317) | -4.38 (0.321)
  Depression Scale at Week 1 (n=139, 137, 138, 137) | -0.32 (0.217) | -0.90 (0.217) | -0.74 (0.216) | -0.92 (0.218)
  Depression Scale at Week 4 (n=137, 138, 135, 134) | -2.32 (0.348) | -3.45 (0.347) | -3.32 (0.350) | -3.80 (0.352)
  Depression Scale at Week 8 (n=129, 129, 127, 122) | -3.19 (0.392) | -4.67 (0.393) | -5.02 (0.396) | -5.49 (0.401)

18. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Physical Functioning Subscore at All Weeks Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The physical functioning subscale assesses limitations in physical activities because of health problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 2, 4 and 8
Population: Full analysis set with available SF-36 Subscore data at Baseline. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 137 | 136
scores on a scale
  Week 2 (n=138,139,136,136) | 2.24 (1.279) | 5.39 (1.273) | 7.55 (1.285) | 3.34 (1.289)
  Week 4 (n=135,132,135,128) | 5.10 (1.354) | 7.77 (1.364) | 9.35 (1.356) | 6.92 (1.385)
  Week 8 (n=129,129,128,122) | 8.77 (1.407) | 9.59 (1.408) | 12.31 (1.411) | 11.28 (1.441)

19. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Role-Physical Subscore at All Weeks Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The role-physical subscale assesses limitations in usual role activities because of physical health problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 2, 4 and 8
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 137 | 136
scores on a scale
  Week 2 (n=138, 139, 136, 136) | 0.74 (1.511) | 6.09 (1.505) | 7.38 (1.520) | 5.00 (1.525)
  Week 4 (n=135, 132, 135, 128) | 4.53 (1.706) | 10.62 (1.721) | 12.97 (1.709) | 8.28 (1.748)
  Week 8 (n=129, 129, 128, 122) | 8.46 (1.830) | 14.09 (1.833) | 15.64 (1.835) | 15.76 (1.878)

20. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Bodily Pain Subscore at All Weeks Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The bodily pain sub-score scale ranges from 0 (best) - 100 (worst). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 2, 4 and 8
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 137 | 136
scores on a scale
  Week 2 (n=138, 139, 136, 136) | 2.99 (1.630) | 5.06 (1.624) | 4.52 (1.644) | 7.22 (1.644)
  Week 4 (n=135, 132, 135, 128) | 4.45 (1.738) | 5.33 (1.752) | 7.75 (1.744) | 10.66 (1.778)
  Week 8 (n=129, 129, 128, 122) | 7.17 (1.920) | 11.99 (1.920) | 9.63 (1.928) | 12.89 (1.970)

21. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) General Health Subscore at All Weeks Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The general health sub-score scale ranges from 0 (best) - 100 (worst). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 2, 4 and 8
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 137 | 136
scores on a scale
  Week 2 (n=138, 139, 136, 136) | 2.83 (1.048) | 5.54 (1.044) | 5.64 (1.054) | 5.47 (1.056)
  Week 4 (n=135, 132, 135, 128) | 6.51 (1.235) | 8.98 (1.245) | 9.96 (1.238) | 10.99 (1.263)
  Week 8 (n=129, 129, 128, 121) | 8.68 (1.392) | 12.46 (1.395) | 13.67 (1.396) | 13.87 (1.429)

22. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Vitality Subscore at All Weeks Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The vitality sub-score assesses energy and fatigue, and ranges from 0 (best) - 100 (worst). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 2, 4 and 8
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 137 | 136
scores on a scale
  Week 2 (n=138, 139, 136, 136) | 5.97 (1.199) | 10.39 (1.193) | 8.83 (1.205) | 8.03 (1.208)
  Week 4 (n=135, 132, 135, 128) | 12.06 (1.523) | 16.69 (1.536) | 16.04 (1.526) | 16.07 (1.560)
  Week 8 (n=129, 129, 128, 122) | 16.14 (1.748) | 22.34 (1.752) | 21.21 (1.753) | 24.17 (1.793)

23. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Social Functioning Subscore at Other Weeks Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The social functioning subscale assesses limitations in social activities because of physical or emotional problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 2 and 4
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 137 | 136
scores on a scale
  Week 2 (n=138, 139, 136, 136) | 6.38 (1.479) | 9.71 (1.473) | 12.02 (1.486) | 10.03 (1.491)
  Week 4 (n=135, 132, 135, 128) | 12.34 (1.760) | 15.71 (1.775) | 18.57 (1.762) | 15.84 (1.804)
  Week 8 (n=129, 129, 128, 122) | 15.60 (1.989) | 21.71 (1.991) | 21.87 (1.993) | 24.94 (2.040)

24. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Role-Emotional Subscore at All Weeks Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The role-emotional subscale assesses limitations in usual role activities because of emotional problems. The sub-score scale ranges from 0 (best) - 100 (worst). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 2, 4 and 8
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 137 | 136
scores on a scale
  Week 2 (n=138, 139, 136, 136) | 6.84 (1.570) | 8.78 (1.563) | 10.87 (1.579) | 9.93 (1.581)
  Week 4 (n=135, 132, 135, 128) | 12.05 (1.755) | 17.01 (1.772) | 18.08 (1.758) | 14.58 (1.797)
  Week 8 (n=129, 129, 128, 122) | 15.96 (1.941) | 23.06 (1.946) | 22.89 (1.947) | 24.71 (1.990)

25. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Mental Health Subscore at All Weeks Assessed
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The mental health sub-score assesses general mental health (psychological distress and well-being) and ranges from 0 (best) - 100 (worst). LS means are from a mixed model for repeated measurements (MMRM) with Baseline-by-week, center, week, and week-by-treatment as factors in the analysis.
Time Frame: Baseline and Weeks 2, 4 and 8
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 137 | 136
scores on a scale
  Week 2 (n=138, 139, 136, 136) | 6.98 (1.199) | 10.62 (1.192) | 9.56 (1.205) | 10.26 (1.207)
  Week 4 (n= 135, 132, 135, 128) | 13.06 (1.418) | 16.78 (1.429) | 16.56 (1.421) | 16.38 (1.451)
  Week 8 (n=129, 129, 128, 122) | 16.28 (1.625) | 23.61 (1.628) | 22.24 (1.631) | 24.89 (1.667)

26. Secondary Outcome: Healthcare Resource Utilization as Assessed by the Health Economic Assessment Questionnaire.
Description: Healthcare resource utilization was assessed by the Health Economic Assessment (HEA) questionnaire, which monitors the participants' absenteeism from work, as well as resource use such as visits to a general practitioner, outpatient and inpatient services, hospitalization, medications, and other relevant services over the past 8 weeks.
Time Frame: Baseline and Week 8
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Number analyzed (Participants) | 139 | 139 | 139 | 139
participants
  Baseline: Any resource use | 62 | 64 | 71 | 61
  Baseline: Any hospitalization-related services | 4 | 3 | 6 | 4
  Baseline: Hospitalization related to depression | 3 | 3 | 4 | 2
  Baseline: Any sick leave | 17 | 7 | 14 | 21
  Baseline: Sick leave related to depression | 12 | 6 | 10 | 18
  Week 8: Any resource use | 31 | 13 | 25 | 25
  Week 8: Any hospitalization-related service | 3 | 0 | 1 | 2
  Week 8: Hospitalization related to depression | 0 | 0 | 1 | 0
  Week 8: Any sick leave | 16 | 6 | 11 | 18
  Week 8: Sick leave related to depression | 13 | 6 | 9 | 14

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are defined as adverse events whose onset occurred or intensity increased after the first dose of double-blind study drug through 30 days after permanent discontinuation of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vortioxetine 1 mg | Vortioxetine 5 mg | Vortioxetine 10 mg
Serious Adverse Events (participants affected / at risk) | 2/140 | 1/140 | 1/140 | 2/139
Other Adverse Events (participants affected / at risk) | 39/140 | 36/140 | 56/140 | 39/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=140) | Vortioxetine 1 mg (N=140) | Vortioxetine 5 mg (N=140) | Vortioxetine 10 mg (N=139)
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=140) | Vortioxetine 1 mg (N=140) | Vortioxetine 5 mg (N=140) | Vortioxetine 10 mg (N=139)
Tachycardia (Cardiac disorders) | 3 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 3 | 4 | 3
Nausea (Gastrointestinal disorders) | 6 | 11 | 22 | 18
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3 | 4
Dry mouth (Gastrointestinal disorders) | 3 | 2 | 3 | 3
Constipation (Gastrointestinal disorders) | 1 | 2 | 3 | 1
Fatigue (General disorders) | 0 | 3 | 5 | 1
Nasopharyngitis (Infections and infestations) | 8 | 5 | 7 | 3
Influenza (Infections and infestations) | 2 | 2 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3 | 1
Headache (Nervous system disorders) | 11 | 9 | 16 | 7
Dizziness (Nervous system disorders) | 3 | 1 | 5 | 9
Somnolence (Nervous system disorders) | 2 | 1 | 3 | 3
Sedation (Nervous system disorders) | 0 | 0 | 3 | 0
Restlessness (Psychiatric disorders) | 1 | 1 | 3 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 2
Hypertension (Vascular disorders) | 3 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.